CLINICAL TRIAL: NCT02080741
Title: Study in Leucocytes From Patients With Type 1 and Type 2 Diabetes Genetic Markers of Inflammation and Oxidative Stress (TÉLOMÈRES/ CANDIDATE GENES) According to the Type A or Type B Behavior Profile
Acronym: Diatolepsy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of inclusion
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CHAUVET-GELINIER APJ 2013
Record Dates: First submitted 2014-03-05; First posted 2014-03-06 (Estimated); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Patients With Type 1 or Type 2 Diabetes; Patients With a Type A or B Behaviour Profile
MeSH Terms: conditions — Diabetes Mellitus, Type 2

ARMS (2):
- Type A behaviour profile (Other)
  Interventions: Other: Blood sample of 12 ml
- Type B behaviour profile (Other)
  Interventions: Other: Blood sample of 12 ml

INTERVENTIONS:
Other: Blood sample of 12 ml

SUMMARY:
This study will include 100 patients with Type 1 and Type 2 diabetes, split into 2 groups of 50 patients according to their behaviour type, and their adaptation to different factors of stress encountered in their lives:

* the first group will consist of patients with a characteristic Type A behaviour profile, that is to say patients with a "proactive, impatient" behaviour pattern
* the second group will consist of patients with a characteristic Type B behaviour profile that is to say patients with a "calm, slow" behaviour pattern The objective is to know if the different behaviour patterns are associated with distinct biological markers likely to influence the evolution of the diabetes.

Participation in this study will be approximately 1h30, patients will participate ONCE ONLY:

1. they will answer simple questions about their disease and then complete 3 questionnaires each with 14 items.
2. they will meet a clinical psychologist for an interview lasting approximately 45 minutes recorded on an audio recorder. The consultation will be used to seek links between the psyche and the disease.
3. they will provide one blood sample of 12 ml (equivalent to a soup spoon) drawn in the morning.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have provided written informed consent
* Patients with type 1 or type 2 diabetes
* Patient admitted for a consultation, as out or in-patients to the Endocrinology-Diabetology-Metabolic diseases department of Dijon CHU
* Patient > 18 years
* Patient with either a characteristic Type A behaviour profile (Bortner > 210), or a characteristic Type B behaviour profile (Bortner<154)

Exclusion Criteria:

* Persons not covered by national health insurance
* Adults under guardianship or wards of court or not intellectually independent
* Patients without diabetes
* Patients with a mixed A/B behaviour profile (154< Bortner score <210)
* Pregnant or breast-feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2014-09-23 (Actual); Primary Completion 2018-05-29 (Actual)

PRIMARY OUTCOMES:
Telomere length | Baselines

SECONDARY OUTCOMES:
Level of expression of candidate genes | Baselines

OTHER OUTCOMES:
Complications of diabetes (Nephropathy, Retinopathy, Neuropathy, Coronaropathy) | Baselines
Scores on psychiatric/psychological scales | Baselines
Analysis of the specific psychological interview EMIC | Baselines

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de DIJON, Dijon, France

REFERENCES:
- [Result] Chauvet-Gelinier JC, Mosca-Boidron AL, Lemogne C, Ragot S, Forestier N, Callegarin D, Allard C, Rebai A, Bouillet B, Ponavoy E, Simoneau I, Petit JM, Bondolfi G, Callier P, Trojak B, Bonin B, Verges B. Type A competitiveness traits correlate with downregulation of c-Fos expression in patients with type 1 diabetes. Diabetes Metab. 2019 Dec;45(6):582-585. doi: 10.1016/j.diabet.2018.11.005. Epub 2018 Nov 23. PMID 30476653